CLINICAL TRIAL: NCT04261972
Title: Early Detection of Cancer in High-risk Patients Through Cell-free DNA 1
Brief Title: Cell-free DNA in Hereditary And High-Risk Malignancies 1
Acronym: CHARM1
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sinai Health System (Other); Women's College Hospital (Other); Jewish General Hospital (Other); IWK Health Centre (Other); British Columbia Cancer Agency (Other); Eastern Health (Other)
Responsible Party: Sponsor
Other Study IDs: 1655
Record Dates: First submitted 2020-01-02; First posted 2020-02-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Cancer Syndrome
Keywords: Circulating tumour DNA; Cell-free DNA (cfDNA); Hereditary cancer syndrome; Cancer; BRCA1; Lynch syndrome; Hereditary breast and ovarian cancer; Liquid biopsies; BRCA2
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary Breast and Ovarian Cancer Syndrome | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Longitudinal blood plasma collected annually on patients. Archived formalin-fixed paraffin-embedded tissue or fresh frozen tissue from a biopsy or surgery is collected when applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHARM: Patients identified with hereditary breast and ovarian cancer syndrome (germline BRCA1 or BRCA2 carrier) or Lynch syndrome (germline variant in EPCAM, MLH1, MSH2, MSH6, or PMS2).
  Interventions: Genetic: Next generation sequencing (NGS)

INTERVENTIONS:
Genetic: Next generation sequencing (NGS) — NGS

SUMMARY:
The goal of this study is to develop an effective, sensitive blood test that can detect early tumours in patients with known or suspected hereditary cancer syndromes (HCS). If this new blood test is accurate, it could be used to screen patients for cancer and allow for earlier cancer detection. The study will also use questionnaires and interviews to understand how patients feel about incorporating these tests into routine medical care, and the perceptions of the medical value of test results.

DETAILED DESCRIPTION:
The objective of this protocol is to develop a method to detect early signs of cancer in 'previvors' (people with HCS that do not yet have a cancer diagnosis). This will enable prediction of cancer onset so that patients and their doctors can make decisions to treat or prevent the cancers. HCS patients will be recruited from across Canada to provide blood samples before and after cancer diagnosis. In parallel, there will be development of a circulating tumour DNA (ctDNA) -based test to detect early stage cancer and evaluation on the cost-effectiveness and feasibility of integrating such screening protocols into routine clinical care. In concert, consultation with patients and health care providers will occur to create recommendations for use within clinical care.

CHARM1 leads into its follow-up study, CHARM2.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with any known or suspected hereditary cancer predisposition (i.e. individuals with an identified pathogenic or likely pathogenic variant in a cancer predisposition gene and/or a family history of cancer without an identified gene mutation) at any stage in their cancer journey (ie: cancer survivor, unaffected with cancer, current cancer patient).
2. Individual must be greater than 18 years of age
3. Individual must speak English or French to participate in the qualitative interview and/or survey

Exclusion Criteria:

1. Individuals that do not meet the outlined inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be studied includes:
  1. Any individual that underwent clinical genetic testing for hereditary breast and ovarian cancer syndrome or Lynch Syndrome and was found to carry a detectable variant that is likely pathogenic or pathogenic.
  2. Any individual with a suspected cancer predisposition that has not yet received genetic testing.
  3. Any individual who received negative genetic test results but has a strong personal or family history of cancer.
Sampling Method: Probability Sample
Enrollment: 1416 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of biospecimens from 1500 HSC carriers. | up to 4 years
  Facilitate and streamline the collection, banking, and annotation of plasma samples and tumour tissue (if applicable) across Canada.
Collection of clinical data from 1500 HSC carriers. | up to 4 years
  Extract clinical data for all study participants from electronic medical records. Data collection will include family history and medical history.
Detection of early stage cancer in HCS patients using cfDNA. | up to 4 years
  Detect concentration of cfDNA circulating in the blood by shallow whole-genome sequencing, targeted panel analysis, and cfMeDIP.
Evaluation of the clinical utility of a cfDNA test for HSC patients. | up to 4 years
  Conduct qualitative interviews with healthcare providers and patients.
Evaluation of the optimal implementation of cfDNA in clinical practice. | up to 4 years
  Conduct a discrete choice experiment survey with HCS patient and providers.
Evaluation of cfDNA test implementation through cost-effectiveness analysis of cfDNA versus standard of care. | up to 4 years
  Conduct economic modelling using the economic evaluation guidelines from the Canadian Agency for Drugs and Technologies in Health.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kim, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (7):
- Canada (7):
  - BC Cancer Agency, Vancouver, British Columbia
  - Eastern Health, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Sinai Health System, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided